CLINICAL TRIAL: NCT00005199
Title: Balloon Valvuloplasty Registry
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1078
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-05

CONDITIONS: Heart Diseases; Mitral Valve Stenosis; Aortic Valve Stenosis
MeSH Terms: conditions — Heart Diseases; Mitral Valve Stenosis; Aortic Valve Stenosis

SUMMARY:
To establish a registry in order to collect and analyze baseline and outcome data on patients with severe valvular stenosis treated with balloon valvuloplasty.

DETAILED DESCRIPTION:
BACKGROUND:

Valvular stenosis or incompetence results in an estimated 41,000 valve replacements in the United States each year. These replacements are equally distributed between the aortic and mitral valves. An estimated 60 percent of aortic valve replacements are the result of valve stenosis; 20-30 percent of mitral valve replacements are due to stenosis. The risk of operative mortality in single valve replacement ranges from 3 percent to as high as 15 percent depending upon patient characteristics. Morbidity associated with open heart procedures includes wound infection, reoperation for bleeding, and post-operative pain. Most patients with artificial valves require anticoagulant therapy for the rest of their lives and thus face the competing risks of hemorrhage and valve thrombosis/embolism. In addition, there are a number of patients with aortic stenosis who are not candidates for aortic valve replacement because of unacceptable operative risks who might be dramatically improved by balloon valvuloplasty.

The pathophysiologic processes underlying valvular stenosis at the aortic and mitral positions are quite different. Mitral stenosis is an outcome of rheumatic fever. Rheumatic fever is quite unusual in this country but it and its sequelae, rheumatic valvular disease, persist as major public health problems in the Third World. Aortic stenosis is most commonly the result of calcific degeneration of a normal tricuspid aortic valve in the elderly or the result of rheumatic fever but can also develop in a congenital bicuspid aortic valve which becomes progressively more stenotic with age and the wear of abnormal flow patterns.

The results of surgical valvuloplasty differ for mitral and aortic valves. Surgical valvuloplasty (commissurotomy) for mitral stenosis is currently a well-established and commonly used treatment for symptomatic patients with mitral stenosis. Similar attempts at repair of aortic stenosis have been largely unsuccessful. Surgical valvuloplasty for aortic stenosis has, for this reason, been abandoned in favor of valve replacement. Initial attempts at aortic balloon valvuloplasty were, therefore, undertaken in patients who were not surgical candidates; these initial efforts in a small number of patients, coming as they did in the wake of abandoned surgical attempts, were surprisingly successful in reducing gradients and increasing valve area without complications such as embolism or significant regurgitation.

Balloon valvuloplasty began with pediatric cardiologists using catheters designed for dilatation of peripheral arterial stenosis in children with pulmonic stenosis and those with coarctation of the aorta. Balloon dilatation has been quite successful with pulmonic stenosis, and is now an accepted therapeutic maneuver. It is less successful with coarctation of the aorta. As a direct outgrowth of this research, investigators have applied this procedure to mitral and aortic stenosis in adults.

Balloon valvuloplasty is performed in the cardiac catheterization laboratory without general anesthesia. A balloon catheter is inserted percutaneously in the venous side of the circulation and is placed across the mitral valve after puncture of the atrial septum. Inflation of appropriately sized balloons has resulted in marked reduction of transvalvular gradients and increase in calculated valve area in most of the cases thus far reported. Given the success of closed commissurotomy, these are not surprising findings.

A similar procedure has been used in severely stenotic aortic valves by either advancing the balloon through the mitral valve into the aortic position or approaching the valve retrograde. Aortic balloon valvuloplasty has thus far been employed largely in severely ill, elderly patients who are judged not able to tolerate valve replacement. As noted above, results have been quite promising; low mortality and morbidity, substantial hemodynamic improvement and short hospital stays have been observed. These anecdotal reports have led to the application of balloon valvuloplasty in increasing numbers of patients. Major issues needed to be addressed prior to general acceptance of this therapy for both aortic and mitral stenosis and for operative and nonoperative candidates. The issues include: definition of risk of mortality and morbidity overall and in subgroups defined by baseline characteristics; success rate defined clinically and hemodynamically overall and in subgroups; the durability of this procedure, that is, how long will a given improvement in clinical and hemodynamic measures persist; definition of subgroups with particularly favorable or unfavorable outcomes. These questions were addressed by the NHLBI Balloon Valvuloplasty Registry.

DESIGN NARRATIVE:

Investigators treating patients with balloon valvuloplasty voluntarily collected and submitted data on consecutive cases of valvuloplasty for two years of active recruitment and followed patients at selected intervals for a minimum of two and a half years. Demographic, clinical, and hemodynamic data were collected on each patient during the valvuloplasty hospitalization. The data were submitted from the participating clinical units to the Coordinating Center.

ELIGIBILITY:
No eligibility criteria

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1987-06; Study Completion 1994-11

REFERENCES:
- [Background] Reid CL, Otto CM, Davis KB, Labovitz A, Kisslo KB, McKay CR. Influence of mitral valve morphology on mitral balloon commissurotomy: immediate and six-month results from the NHLBI Balloon Valvuloplasty Registry. Am Heart J. 1992 Sep;124(3):657-65. doi: 10.1016/0002-8703(92)90274-y. PMID 1514494
- [Background] Davidson CJ, Bashore TM, Mickel M, Davis K. Balloon mitral commissurotomy after previous surgical commissurotomy. The National Heart, Lung, and Blood Institute Balloon Valvuloplasty Registry participants. Circulation. 1992 Jul;86(1):91-9. doi: 10.1161/01.cir.86.1.91. PMID 1617794
- [Background] Otto CM, Davis KB, Holmes DR Jr, O'Neill W, Ferguson J, Bashore TM, Bonan R. Methodologic issues in clinical evaluation of stenosis severity in adults undergoing aortic or mitral balloon valvuloplasty. The NHLBI Balloon Valvuloplasty Registry. Am J Cardiol. 1992 Jun 15;69(19):1607-16. doi: 10.1016/0002-9149(92)90712-8. PMID 1598878
- [Background] Complications and mortality of percutaneous balloon mitral commissurotomy. A report from the National Heart, Lung, and Blood Institute Balloon Valvuloplasty Registry. Circulation. 1992 Jun;85(6):2014-24. doi: 10.1161/01.cir.85.6.2014. PMID 1591821
- [Background] Multicenter experience with balloon mitral commissurotomy. NHLBI Balloon Valvuloplasty Registry Report on immediate and 30-day follow-up results. The National Heart, Lung, and Blood Institute Balloon Valvuloplasty Registry Participants. Circulation. 1992 Feb;85(2):448-61. doi: 10.1161/01.cir.85.2.448. PMID 1735143
- [Background] Otto CM, Nishimura RA, Davis KB, Kisslo KB, Bashore TM. Doppler echocardiographic findings in adults with severe symptomatic valvular aortic stenosis. Balloon Valvuloplasty Registry Echocardiographers. Am J Cardiol. 1991 Dec 1;68(15):1477-84. doi: 10.1016/0002-9149(91)90282-p. PMID 1746430
- [Background] Percutaneous balloon aortic valvuloplasty. Acute and 30-day follow-up results in 674 patients from the NHLBI Balloon Valvuloplasty Registry. Circulation. 1991 Dec;84(6):2383-97. doi: 10.1161/01.cir.84.6.2383. PMID 1959194
- [Background] Otto CM, Mickel MC, Kennedy JW, Alderman EL, Bashore TM, Block PC, Brinker JA, Diver D, Ferguson J, Holmes DR Jr, et al. Three-year outcome after balloon aortic valvuloplasty. Insights into prognosis of valvular aortic stenosis. Circulation. 1994 Feb;89(2):642-50. doi: 10.1161/01.cir.89.2.642. PMID 8313553
- [Background] Otto CM, Davis KB, Reid CL, Slater JN, Kronzon I, Kisslo KB, Bashore TM. Relation between pulmonary artery pressure and mitral stenosis severity in patients undergoing balloon mitral commissurotomy. Am J Cardiol. 1993 Apr 1;71(10):874-8. doi: 10.1016/0002-9149(93)90844-3. No abstract available. PMID 8456774
- [Background] Douglas PS, Otto CM, Mickel MC, Labovitz A, Reid CL, Davis KB. Gender differences in left ventricle geometry and function in patients undergoing balloon dilatation of the aortic valve for isolated aortic stenosis. NHLBI Balloon Valvuloplasty Registry. Br Heart J. 1995 Jun;73(6):548-54. doi: 10.1136/hrt.73.6.548. PMID 7626355
- [Background] Engbaek F, Voldby B. Radioimmunoassay of serotonin (5-hydroxytryptamine) in cerebrospinal fluid, plasma, and serum. Clin Chem. 1982 Apr;28(4 Pt 1):624-8. PMID 7074830